CLINICAL TRIAL: NCT01399229
Title: Comparison of SureCALL® Labor Monitor® and Tocodynamometer Measurement in Preterm and Term Pregnant Women
Status: Completed | Type: Observational
Sponsor: Reproductive Research Technologies, LP (Industry)
Responsible Party: Sponsor
Other Study IDs: RRT-11-01
Record Dates: First submitted 2011-07-19; First posted 2011-07-21 (Estimated); Results first posted 2013-08-27 (Estimated); Last update posted 2013-09-12 (Estimated); Status verified 2013-08

CONDITIONS: Pregnancy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Pregnant, Preterm, In Labor: Gestation Age at or less than 36 weeks, clinically determined to be in labor
- Pregnant, Preterm, Nonlaboring: Gestation Age at or less than 36 weeks, clinically determined to not be in labor
- Pregnant, Term, Nonlaboring: Gestation Age more than 36 weeks, clinically determined to not be in labor

SUMMARY:
This measurement study was designed to evaluate the performance of SureCALL® Labor Monitor® (SureCALL®) compared to the predicate Tocodynamometer device (TOCO) in preterm and term pregnant patients.

DETAILED DESCRIPTION:
The SureCALL® Labor Monitor® (SureCALL®) is a transabdominal electromyography monitor intended to measure uterine activity. It is intended for use on pregnant women, with singleton pregnancies, using surface electrodes on the maternal abdomen. The device is intended for use by healthcare professionals in a clinical setting.

This measurement study was designed to evaluate the performance of SureCALL® Labor Monitor® (SureCALL®) compared to the predicate Tocodynamometer device (TOCO) in pregnant laboring preterm patients, nonlaboring preterm patients, and nonlaboring term patients.

This study involved 25 women at a Gestational Age of 36 weeks or less and 5 women at a Gestation Age of greater than 36 at five clinical sites. Each study subject was instrumented with two technologies for measuring uterine activity:

1. Standard tocodynamometer attached to the maternal abdomen,
2. SureCALL® with a set of abdominal surface electrodes for uterine electromyography attached to the maternal abdomen

Subjects did not recieve any interventions as a part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Singleton Pregnancy
* Informed Consent Required

Exclusion Criteria:

* Multifetal Pregnancy
* Informed Consent Not Given

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women with uncomplicated singleton pregnancies
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2007-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy B Waterhouse, MD, Study Director — Reproductive Research Technologies, LP
Locations (5):
- United States (5):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Southeast Texas OB/GYN Associates, Beaumont, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Woman's Hospital of Texas, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Pregnant, Preterm, In Labor: Pregnant preterm women independently determined to be in labor.
- Pregnant, Preterm, Non Labor: Pregnant preterm women independently determined to not be in labor.
- Pregnant, Term, Non Labor: Pregnant term women independently determined to be in labor.
Period: Overall Study
Arm/Group | Pregnant, Preterm, In Labor | Pregnant, Preterm, Non Labor | Pregnant, Term, Non Labor
Started | 20 | 5 | 5
Completed | 20 | 5 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pregnant: The study focused on recruiting laboring preterm patients, nonlaboring preterm patients, and nonlaboring term patients.
Arm/Group | Pregnant
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 28
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 29.50 (6.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Comparison of SureCALL® and Tocodynamometer Detection of Contraction Event Timing
Description: Time Stamps of the Peaks of Corresponding Contractions
Time Frame: 9 - 41 Minutes
Measure: Mean (Standard Deviation); unit: Seconds
Groups:
- Pregnant Patents With Uterine Contractions: Patient contractions were monitored with both SureCALL® Labor Monitor® and Tocodynamometer. The times of peak contractions recorded by both devices were compared, and the time differences between contractions were assessed.
Arm/Group | Pregnant Patents With Uterine Contractions
Number analyzed (Participants) | 30
Seconds | 0.99 (15.17)
Statistical Analysis 1: Comparison: Pregnant Patents With Uterine Contractions; Test type: Non-Inferiority or Equivalence — Agreement between SureCALL® and Tocodynamometer Contraction Peak Times Null hypothesis: The mean peak difference between RMS and TOCO is equal to 0. Alternative hypothesis: The mean peak difference is not equal to 0; p = 0.4901, Mixed Models Analysis; Mean Difference (Net) = .99, 95% CI 2-sided [-28.74 to 30.72], Standard Error of Mean 1.4086

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the date of each patient's enrollment through delivery.
Description: There were no interventions as a part of the study and no adverse events related to the study reported.
Arm/Group | Pregnant
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs may publish or present results of the study after the expiration of 12 months from completion. Publications or presentations are subject to the protection of confidential information or patentable information.